CLINICAL TRIAL: NCT07354841
Title: A Two Phases Clinical Investigation Consisting of a Pre-Market, Pilot, Interventional, Not Randomized, Monocentric Investigation to Evaluate the Safety of PVC Arterial Cannula and PVC Venous Cannula (Class III Medical Devices) Intended to be Used During Cardiopulmonary Bypass (CPB) Procedure Followed by a Pre-Market, Pivotal, Interventional, Randomized, Non- Inferiority, Monocentric Investigation to Confirm the Safety and Evaluate the Performance of the Same Cannulas
Brief Title: Safety and Performance Evaluation of CPB Venous and Arterial Cannulas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eurosets S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: DE-62-22; CIV-IT-25-03-051856 (Other: Eudamed)
Record Dates: First submitted 2025-11-20; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Surgery; Heart Surgery; Cardiopulmonary Bypass; Coronary Surgery; Aortic Valve Surgery; Cannulation; Venous Cannulation; Arterial Cannulation; Coronary Surgery With Cardiopulmonary Bypass
Keywords: Arterial Cannula; Venous Cannula; Extracorporeal Circulation; Cardiopulmonary Bypass; Cardiac Surgery; Medical Device; Device Safety; Device Performance; Aortic Valve Surgery; Coronary Surgery; Two Phases clinical investigation; Monocentric Study; Two Phases Study; Serious Adverse Events (SAE); CVP; NIRS; Venous Cannula Drainage Pressure; Arterial Cannula Reinfusion Pressure

STUDY DESIGN:
Intervention Model Description: Phase 1: Pilot, not Randomized, Monocentric one arm Clinical Investigation with pre-market medical device Phase 2: Pivotal, Randomized, Non-inferiority, Monocentric, two arm Clinical Investigation with pre-market medical device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eurosets Arterial and Venous Cannula (Experimental): Phase 1: All enrolled subjects will undergo cardiopulmonary bypass using the investigational Eurosets arterial and venous cannulas to evaluate the safety.
  Phase 2: Participants will undergo cardiopulmonary bypass using the investigational Eurosets arterial and venous cannulas to confirm safety and to evaluate the performance.
  Interventions: Device: Eurosets Venous and Arterial Cannula
- Control Arterial and Venous Cannula (Active Comparator): Phase 2: Participants will undergo cardiopulmonary bypass using commercially available arterial and venous cannulas currently used in standard clinical practice.
  Interventions: Device: Control Arterial and Venous Cannulas

INTERVENTIONS:
Device: Eurosets Venous and Arterial Cannula — Phase 1: Use of investigational Eurosets arterial and venous cannulas during CPB to assess safety and preliminary performance.The Arterial cannulae are designed for insertion in the ascending Aorta. For this Investigation the arterial cannula is reinforced-long curved with flange tip, 3/8" connector with luer lock, 24 Fr.The Venous Cannulae are designed to be used for vena cava and right atrium blood drainage during CPB surgery. For this Investigation the venous cannula is dual stage without connector, lighthouse tip, 32/40 Fr.
  Phase 2: Use of investigational PVC arterial and venous cannulas during cardiopulmonary bypass (CPB) to confirm safety and evaluate performance compared to control group. For Investigation device: same of phase 1. For Control Group: the Arterial Cannula is EOPA (Medtronic), 24 Fr; the Venous Cannula is Two stage MC2 (Medtronic), 32/40 Fr.
  Arms: Eurosets Arterial and Venous Cannula
Device: Control Arterial and Venous Cannulas — Phase 2: Use of commercially available arterial and venous cannulas as comparator devices to evaluate the performance of the investigational PVC Arterial and Venous Cannulas during cardiopulmonary bypass (CPB) procedures. the control cannulas are EOPA 24Fr (Medtronic) as Arterial Cannula and Two Stage MC2 32/40Fr (Medtronic) as Venous Cannula.
  Arms: Control Arterial and Venous Cannula

SUMMARY:
This is a two-phase study evaluating the Eurosets arterial and venous cannulas for use during cardiopulmonary bypass (CPB) procedures. Phase 1 is a pilot study focused on assessing cannula safety. Phase 2 is a pivotal study aimed at confirming safety and evaluating efficacy through comparison with Medtronic cannulas (control group).

The results will be compared for non-inferiority with those obtained using the control group cannulas.

DETAILED DESCRIPTION:
The Clinical Investigation is a Two Phases clinical investigation consisting of a pre-Market, Pilot, Interventional, not Randomized, Monocentric Investigation to Evaluate the Safety of PVC Arterial Cannula and PVC Venous Cannula (Class III Medical Devices) intended to be used during Cardiopulmonary Bypass (CPB) procedure followed by a pre-Market, Pivotal, Interventional, Randomized, Non- inferiority, Monocentric Investigation to confirm the Safety and evaluate the Performance of the same cannulas.

The aim of these investigations are: 1) to evaluate safety of Eurosets Venous Cannula and Arterial Cannula in patients subjected to CPB and 2) to evaluate the performance and safety of Arterial Cannula and Venous Cannula intended to be used during CPB procedure. The results obtained will be compared by non-inferiority to the results obtained by Medtronic cannulae (control group).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is considered able and willing to provide written informed consent according to the ethically approved informed consent form;
2. Female and male patients aged ≥ 18;
3. Body weight between 60 and 120 kg;
4. Body surface area (BSA) between 1.5 and 2.5 m2;
5. Patients scheduled to undergo central cannulation for cardiopulmonary bypass (CPB) in elective surgery procedures (isolated coronary and/or aortic valve surgery).

Exclusion Criteria:

1. Emergency cases;
2. Re-do cardiac surgery procedure;
3. Diabetes mellitus;
4. Hematologic diseases or history of thrombophilia;
5. Pregnancy or breastfeeding;
6. Concomitant major cardiac procedures;
7. Active malignant/metastatic neoplasm of any type;
8. Presence of pneumothorax and/or pulmonary emphysema;
9. Significant central nervous system injury;
10. Current intracranial hemorrhage;
11. Immunosuppression;
12. Contraindication for therapeutic anticoagulation (e.g., heparin);
13. Anatomical and structural abnormalities which, in the opinion of the Investigator, may interfere with the participation to the study;
14. Abnormal or pathological cannulation site;
15. Uncontrolled active bleeding;
16. Awaiting transplantation;
17. Requiring preoperative extracorporeal membrane oxygenation;
18. Presence of any relevant severe condition or clinically relevant abnormal laboratory parameters that in the opinion of the Investigator may interfere with the participation to the study.
19. Patient is taking part in another interventional clinical study;
20. Patient is not able to understand the nature of this study or is unwilling or unable to attend the EOS Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Safety of Eurosets Arterial and Venous Cannulas | At Visit 1 (Pre and during surgical procedure), at Visit 2 (24 hours post-surgical procedure) and at Visit 3 (within 6-7 days post-surgical procedure)
  Number and type of adverse events over the duration of the investigation.
Phase 2: Performance of Eurosets Arterial Cannulas | Time points during CPB: 1st: pre-clamping/CPB initiation, 2nd: pre-weaning
  For Arterial cannula: the performance of the Eurosets Arterial Cannulacerebral oximetry (rSO2) will be monitored during CPB using near infrared spectroscopy (NIRS). Delta rSO2 (will be calculated as the percentage) (rate of decrease of rSO2 from pre-clamping) will be compared to delta rSO2 of control arterial cannula.
Phase 2: Performance of Eurosets Venous Cannulas | Time points during CPB: 1st: pre-clamping/CPB initiation (full flow), 2nd: 10 minutes post-clamping, 3rd: 30 minutes post-clamping.
  For Venous cannula: the performance of the Eurosets Venous Cannula, Central Venous Pressure (CVP) values will be monitored during CPB. Results will be compared to control venous cannula.

SECONDARY OUTCOMES:
Phase 1: Clinical Parameters collected for safety: pH | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Clinical parameters monitored with pH value
Phase 1: Clinical Parameters collected for safety: pCO2 | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Clinical parameters: pCO2 recorded with mmHg
Phase 1: Clinical Parameters collected for safety: pO2 | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Clinical parameters: pO2 recorded with mmHg
Phase 1: Clinical Parameters collected for safety: Blood Flow | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Clinical parameters: Blood flow recorded with L/min
Phase 1: Clinical Parameters collected for safety: Mean arterial pressure (MAP) | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Clinical parameters: MAP recorded with mmHg
Phase 1: Clinical Parameters collected for safety: Mixed venous oxygen saturation (SvO2) | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Clinical parameters: SvO2 recorded with percentage (%)
Phase 1: Clinical Parameters collected for safety: Arterial oxygen saturation (SaO2) | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Clinical parameters: SaO2 monitored with percentage
Phase 1: Clinical Parameters collected for safety: Vacuum level | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Clinical parameters: Vacuum level monitored with mmHg
Phase 1: Vital sign collected for safety: body temperature | At Visit 0 (from day -3 to day -1), Day of Surgery - Visit 1 (Day 0), Visit 2 (24 hours after surgery), Visit 3 (6-7 days after surgery), at Unscheduled Visit(s).
  Vital signs: Body Temperature recorded with Celsius degrees (T°)
Phase 1: Vital sign collected for safety: Heart Rate | At Visit 0 (from day -3 to day -1), Day of Surgery - Visit 1 (Day 0), Visit 2 (24 hours after surgery), Visit 3 (6-7 days after surgery).
  Vital signs: Heart Rate recorded with beats/min
Phase 1: Vital Sign collected for safety: Blood Flow | At Visit 0 (from day -3 to day -1), Day of Surgery - Visit 1 (Day 0), Visit 2 (24 hours after surgery), Visit 3 (6-7 days after surgery).
  Vital Sign: Blood flow recorded with L/min
Phase 1: Vital sign collected for safety: Diastolic pressure | At Visit 0 (from day -3 to day -1), Day of Surgery - Visit 1 (Day 0), Visit 2 (24 hours after surgery), Visit 3 (6-7 days after surgery).
  Vital signs: Diastolic pressure recorded with mmHg
Phase 1: Vital sign collected for safety: Sistolic pressure | At Visit 0 (from day -3 to day -1), Day of Surgery - Visit 1 (Day 0), Visit 2 (24 hours after surgery), Visit 3 (6-7 days after surgery).
  Vital signs: Sistolic pressure recorded with mmHg
Phase 1: Vital sign collected for safety: SpO2 | At Visit 0 (from day -3 to day -1), Day of Surgery - Visit 1 (Day 0), Visit 2 (24 hours after surgery), Visit 3 (6-7 days after surgery).
  Vital signs: SpO2 recorded with percentage (%)
Phase 1: Device deficiencies/incidents collected for safety | At Visit 1 Day 1 (Day of surgery): pre-CPB; 1st time point: Pre-clamping/CPB initiation; 2nd time point: 10 minutes post-clamping; 3rd time point: 30 minutes post-clamping; (pre) weaning/decannulation.
  Device deficiencies/incidents: recorded with number of Device Deficiencies or Incidents
Phase 1: Concomitant medications collected for safety | At Visit 0 (from day -3 to day -1), Day of Surgery - Visit 1 (Day 0), Visit 2 (24 hours after surgery), Visit 3 (6-7 days after surgery).
  Concomitant medications: Medications administered (dosage) during the study period.
Phase 1: Drainage pressure collected for safety | At visit 1 Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping.
  Drainage pressure: venous pressure compared to blood flow recorded with mmHg
Phase 1: Reinfusion pressure collected for safety | At visit 1 Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping.
  Reinfusion pressure: arterial pressure compared to blood flow recorded with mmHg
Phase 1: Adequacy of tissue perfusion collected for safety | At Visit 1 Day 1 (Day of surgery): (pre) weaning/ decannulation
  Adequacy of tissue perfusion recorded with levels of blood lactate
Phase 1: Patient's metabolic condition collected for safety: indexed oxygen delivery (DO2i ) | At visit 1 Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Patient's metabolic condition DO2i recorded with ml/min/m2
Phase 1: Patient's metabolic condition collected for safety: oxygen consuption (VO2) | At visit 1 Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Patient's metabolic condition VO2 recorded with ml/min
Phase 1: Patient's metabolic condition collected for safety: oxygen extraction (O2ER) | At visit 1 Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Patient's metabolic condition O2ER recorded with percentage (%)
Phase 1: Patient's metabolic condition collected for safety: venous oxygen saturation (SvO2) | At visit 1 Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Patient's metabolic condition SvO2 recorded with percentage (%)
Phase 1: Patient's metabolic condition coillected for safety: arterial oxygen saturation (SaO2) | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Patient's metabolic condition SaO2 recorded with percentage (%)
Phase 1: Drainage efficacy of the venous cannula collected for safety | At Visit 0 (from day -3 to day -1 of surgical procedure) and Visit 2 (24 hours post-surgical procedure)
  Drainage efficacy of the venous cannula recorded with levels of bilirubin
Phase 1: Drainage efficacy of the venous cannula collected for safety | At Visit 0 (from day -3 to day -1 of surgical procedure) and Visit 2 (24 hours post-surgical procedure)
  Drainage efficacy of the venous cannula recorded with levels of creatinine
Phase 1: Drainage efficacy of the venous cannula collected for safety | At Visit 0 (from day -3 to day -1 of surgical procedure) and Visit 2 (24 hours post-surgical procedure)
  Drainage efficacy of the venous cannula recorded with levels of transaminases
Phase 1: Duration of CPB procedure and clamping collected for safety | At Visit 1 Day 1 (day of surgery): (pre) weaning/ decannulation.
  Duration of CPB procedure and clamping recorded with Time (minutes)
Phase 1: (de)cannulation difficulty collected for safety | At Visit 1 Day 1 (day of surgery): (pre) weaning/ decannulation
  (de)cannulation difficulty recorded with 5-likert Scale (from 1 - very easy to 5 - very difficult) completed by the anesthesiologist/perfusionist/physician who performed the procedure at Visit 1.
Phase 1: Integrity of arterial and venous cannula at decannulation collected for safety | At Visit 1 Day 1 (day of surgery): (pre) weaning/ decannulation
  Integrity of arterial and venous cannula at decannulation will be evaluated by the anesthesiologist/perfusionist/physician who performed the procedure and recorded with YES or NO.
Phase 1: Presence of clots or thrombi in arterial and venous cannula at decannulation collected for safety | At Visit 1 Day 1 (day of surgery): (pre) weaning/ decannulation
  Presence of clots or thrombi in arterial and venous cannula at decannulation. The presence of clots or thrombi will be recorded with YES or NO on the eCRF.
Phase 1: Hospitalization stay collected for safety | At Visit 3: Pre-discharge (within 6-7 days post-surgical procedure)
  The number of hospitalization days will be recorded up to patient discharge.
Phase 2: Drainage pressure (Pdrain) collected for non-inferiority with control group | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Drainage pressure (Pdrain) recorded with mmHg. Results compared with control Venous Cannula.
Phase 2: Reinfusion pressure (Pout) collected for non-inferiority with control group | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Reinfusion pressure recorded with mmHg. Results compared with control Arterial Cannula.
Phase 2: Adequacy of tissue perfusion collected for non-inferiority with control group | At Visit 1. Day 1 (Day of surgery): (pre) weaning/decannulation.
  Adequacy of tissue perfusion recorded with levels of blood lactate. Results compared with control group
Phase 2: Patient's metabolic condition collected for non-inferiority with control group: indexed oxygen delivery (DO2i) | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Patient's metabolic condition DO2i recorded with ml/min/m2. Results compared with control group.
Phase 2: Patient's metabolic condition collected for non-inferiority with control group: oxygen consumption (VO2) | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Patient's metabolic condition VO2 recorded with ml/min. Results compared with control group.
Phase 2: Patient's metabolic condition collected for non-inferiority with control group: oxygen extraction (O2ER) | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Patient's metabolic condition O2ER recorded with percentage (%). Results compared with control group.
Phase 2: Patient's metabolic condition collected for non-inferiority with control group: venous oxygen saturation (SVO2) | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Patient's metabolic condition SVO2 recorded with percentage (%). Results compared with control group.
Phase 2: Patient's metabolic condition collected for non-inferiority with control group: arterial oxygen ssaturation (SaO2) | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Patient's metabolic condition SaO2 recorded with percentage (%). Results compared with control group.
Phase 2: Drainage efficacy of the venous cannula collected for non-inferiority with control group | At screening/baseline (Visit 0): Within 3 days before the day of surgery. At Visit 2: 24 hours post-surgical procedure. At Visit 3: before discharge (6-7 days post-surgical procedure).
  Drainage efficacy of the venous cannula recorded with levels of bilirubin. Results compared with control group.
Phase 2: Drainage efficacy of the venous cannula collected for non-inferiority with control group | At screening/baseline (Visit 0): Within 3 days before the day of surgery. At Visit 2: 24 hours post-surgical procedure. At Visit 3: before discharge (6-7 days post-surgical procedure).
  Drainage efficacy of the venous cannula recorded with levels of creatinine. Results compared with control group.
Phase 2: Drainage efficacy of the venous cannula collected for non-inferiority with control group | At screening/baseline (Visit 0): Within 3 days before the day of surgery. At Visit 2: 24 hours post-CPB. At Visit 3: before discharge (6-7 days post-surgical procedure).
  Drainage efficacy of the venous cannula recorded with levels of transaminases. Results compared with control group.
Phase 2: Duration of CPB procedure and clamping time collected for non-inferiority with control group | At Visit 1. Day 1 (Day of Surgery): (pre) weaning/decannulation.
  Duration of CPB procedure and clamping time recorded with Time (minutes). Results compared with control group.
Phase 2: (de)cannulation difficulty collected for non-inferiority with control group | At Visit 1. Day 1 (Day of Surgery): (pre) weaning/decannulation.
  (de)cannulation difficulty recorded with 5-likert Scale (from 1 - very easy to 5 - very difficult) completed by the anesthesiologist/perfusionist/physician. Results compared with control group.
Phase 2: Integrity of arterial and venous cannula at decannulation collected for non-inferiority with control group | At Visit 1. Day 1 (Day of Surgery): (pre) weaning/decannulation.
  Integrity of arterial and venous cannula at decannulation recorded with YES or NO.
Phase 2: Presence of clots or thrombi in arterial and venous cannula at decannulation collected for non-inferiority with control group | At Visit 1. Day 1 (Day of Surgery): (pre) weaning/decannulation.
  Presence of clots or thrombi in arterial and venous cannula at decannulation recorded with YES or NO on the eCRF. Results compared with control cannulae.
Phase 2: Hospitalization stay collected for non-inferiority with control group | At Visit 3 (End of Study). Pre-discharge (6-7 days post-surgical procedure).
  Hospitalization stay recorded with number of hospitalization days. Results compared with control group

OTHER OUTCOMES:
Safety Endpoint during Phase 2 (Pivotal): Monitoring of clinical parameters: pH | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Clinical parameters monitored with pH value
Safety Endpoint during Phase 2 (Pivotal): Monitoring of clinical parameters: pCO2 | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Clinical parameters: pCO2 recorded with mmHg
Safety Endpoint during Phase 2 (Pivotal): Monitoring of clinical parameters: pO2 | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Clinical parameters: pO2 recorded with mmHg
Safety Endpoint during Phase 2 (Pivotal): Monitoring of clinical parameters: Bloof flow | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Clinical parameters: Blood flow recorded with L/min
Safety Endpoint during Phase 2 (Pivotal): Monitoring of clinical parameters: Mean arterial Pressure (MAP) | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Clinical parameters: MAP recorded with mmHg
Safety Endpoint during Phase 2 (Pivotal): Monitoring of clinical parameters: Mixed venous oxygen saturation (SvO2) | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Clinical parameters: SvO2 recorded with percentage (%)
Safety Endpoint during Phase 2 (Pivotal): Monitoring of clinical parameters: Arterial oxygen saturation (SaO2) | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Clinical parameters: SaO2 monitored with percentage (%)
Safety Endpoint during Phase 2 (Pivotal): Monitoring of clinical parameters: Vaccum Level | At Visit 1. Day 1 (Day of surgery): 1st time point: Pre-clamping/CPB initiation, 2nd time point: 10 minutes post-clamping, 3rd time point: 30 minutes post-clamping, (pre) weaning/ decannulation.
  Clinical parameters: Vacuum level monitored with mmHg
Safety Endpoint during Phase 2 (Pivotal): Monitoring of vital sign: Body temperature | At Visit 0 (from day -3 to day -1), Day of Surgery - Visit 1 (Day 0), Visit 2 (24 hours after surgery), Visit 3 (6-7 days after surgery).
  Description: Vital signs: Body Temperature recorded with Celsius degree (T°)
Safety Endpoint during Phase 2 (Pivotal): Monitoring of vital sign: Heart Rate | At Visit 0 (from day -3 to day -1), Day of Surgery - Visit 1 (Day 0), Visit 2 (24 hours after surgery), Visit 3 (6-7 days after surgery).
  Vital signs: Heart Rate recorded with beats/min
Safety Endpoint during Phase 2 (Pivotal): Monitoring of vital sign: Blood flow | At Visit 0 (from day -3 to day -1), Day of Surgery - Visit 1 (Day 0), Visit 2 (24 hours after surgery), Visit 3 (6-7 days after surgery).
  Vital Sign: Blood flow recorded with L/min
Safety Endpoint during Phase 2 (Pivotal): Monitoring of vital sign: diastolic pressure | At Visit 0 (from day -3 to day -1), Day of Surgery - Visit 1 (Day 0), Visit 2 (24 hours after surgery), Visit 3 (6-7 days after surgery).
  Vital signs: Diastolic pressure recorded with mmHg
Safety Endpoint during Phase 2 (Pivotal): Monitoring of vital sign: sistolic pressure | At Visit 0 (from day -3 to day -1), Day of Surgery - Visit 1 (Day 0), Visit 2 (24 hours after surgery), Visit 3 (6-7 days after surgery).
  Vital signs: Sistolic pressure recorded with mmHg
Safety Endpoint during Phase 2 (Pivotal). Monitoring of vital sign: SpO2 | At Visit 0 (from day -3 to day -1), Day of Surgery - Visit 1 (Day 0), Visit 2 (24 hours after surgery), Visit 3 (6-7 days after surgery).
  Vital signs: SpO2 recorded with percentage (%)
Safety Endpoint during Phase 2 (Pivotal): Monitoring of Device deficiencies/incidents | At Visit 1 Day 1 (Day of surgery): pre-CPB; 1st time point: Pre-clamping/CPB initiation; 2nd time point: 10 minutes post-clamping; 3rd time point: 30 minutes post-clamping; (pre) weaning/decannulation.
  Device deficiencies/incidents recorded with number of Device Deficiencies or Incidents
Safety Endpoint during Phase 2 (Pivotal): Monitoring of adverse events, and serious adverse events unrelated to study device | At Visit 1 (Pre and during surgical procedure), at Visit 2 (24 hours post-surgical procedure) and at Visit 3 (within 6-7 days post-surgical procedure)
  Number and type of adverse events, and serious adverse events unrelated to study device over the duration of the investigation.
Safety Endpoint during Phase 2 (Pivotal): Monitoring of concomitant medications | At Visit 0 (from day -3 to day -1), Day of Surgery - Visit 1 (Day 0), Visit 2 (24 hours after surgery), Visit 3 (6-7 days after surgery).
  Concomitant medications: Medications administered (dosage) during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Anthea Hospital GVM Care & Research, Bari, BA, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ismail A, Semien G, Sharma S, Collier SA, Miskolczi SY. Cardiopulmonary Bypass. 2024 Aug 12. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482190/ PMID 29489210
- [Result] von Segesser LK, Ferrari E, Delay D, Maunz O, Horisberger J, Tozzi P. Routine use of self-expanding venous cannulas for cardiopulmonary bypass: benefits and pitfalls in 100 consecutive cases. Eur J Cardiothorac Surg. 2008 Sep;34(3):635-40. doi: 10.1016/j.ejcts.2008.05.037. Epub 2008 Jul 16. PMID 18635371
- [Result] Sarkar M, Prabhu V. Basics of cardiopulmonary bypass. Indian J Anaesth. 2017 Sep;61(9):760-767. doi: 10.4103/ija.IJA_379_17. PMID 28970635
- [Result] Authors/Task Force Members; Kunst G, Milojevic M, Boer C, De Somer FMJJ, Gudbjartsson T, van den Goor J, Jones TJ, Lomivorotov V, Merkle F, Ranucci M, Puis L, Wahba A; EACTS/EACTA/EBCP Committee Reviewers; Alston P, Fitzgerald D, Nikolic A, Onorati F, Rasmussen BS, Svenmarker S. 2019 EACTS/EACTA/EBCP guidelines on cardiopulmonary bypass in adult cardiac surgery. Br J Anaesth. 2019 Dec;123(6):713-757. doi: 10.1016/j.bja.2019.09.012. Epub 2019 Oct 2. No abstract available. PMID 31585674
- [Result] Lamelas J, Aberle C, Macias AE, Alnajar A. Cannulation Strategies for Minimally Invasive Cardiac Surgery. Innovations (Phila). 2020 May/Jun;15(3):261-269. doi: 10.1177/1556984520911917. Epub 2020 May 21. PMID 32437215
- [Result] Narasaki S, Miyoshi H, Nakamura R, Sumii A, Watanabe T, Otsuki S, Tsutsumi YM. Venous cannula occlusion during cardiopulmonary bypass recognized by ultrasonography of the internal jugular vein. JA Clin Rep. 2022 Apr 12;8(1):29. doi: 10.1186/s40981-022-00519-2. PMID 35412158
- [Result] Wahba A, Milojevic M, Boer C, De Somer FMJJ, Gudbjartsson T, van den Goor J, Jones TJ, Lomivorotov V, Merkle F, Ranucci M, Kunst G, Puis L; EACTS/EACTA/EBCP Committee Reviewers. 2019 EACTS/EACTA/EBCP guidelines on cardiopulmonary bypass in adult cardiac surgery. Eur J Cardiothorac Surg. 2020 Feb 1;57(2):210-251. doi: 10.1093/ejcts/ezz267. No abstract available. PMID 31576396
- See also: [Yichao et al., 2006] Yichao Teng, HaiShu Ding, Qingcheng Gong, Zaishen Jia, Lan Huang, "Monitoring cerebral oxygen saturation during cardiopulmonary bypass using near-infrared spectroscopy: the relationships with body temperature and perfusion rate," J. — https://doi.org/10.1117/1.2187422